CLINICAL TRIAL: NCT04335877
Title: Effectiveness-Implementation Research to Assess the Effect of Prompting the Supply of Zinc/LO-ORS Co-packs Through the Private Sector Coupled With Behavior Change Intervention on the Treatment of Uncomplicated Childhood Diarrhoea in Kenya
Brief Title: Effect of Prompting the Supply of Zinc/LO-ORS Co-packs in the Private Sector Plus BCI on Childhood Diarrhea Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutrition International (Other)
Responsible Party: Principal Investigator, Elijah Mbiti, Senior Program Officer, Nutrition International
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NI-01-2006-ZNIR
Record Dates: First submitted 2020-03-30; First posted 2020-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Diarrhea, Infantile
MeSH Terms: conditions — Diarrhea, Infantile

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Private sector component + modified BCC (Experimental): Private sector component + modified BCC + current standard of care
  Interventions: Other: Private sector component + modified BCC
- Control (No Intervention): Current standard of care + standard BCC

INTERVENTIONS:
Other: Private sector component + modified BCC — Intervention group will be exposed to the private sector component + modified BCC and will receive current standard care
  Arms: Private sector component + modified BCC

SUMMARY:
This study assesses whether prompting the supply of zinc and LO-ORS co-packs in the private sector coupled with behavior change communication (BCC) has an effect on the treatment of uncomplicated childhood diarrhea. In addition the study will evaluate the acceptability, adoption, feasibility and coverage of the intervention model. One group of children and caregivers will receive the current standard of care and will be exposed to standard BCC and the second group will be exposed to the private sector component and to a modified BCC.

DETAILED DESCRIPTION:
Diarrhoea accounts for 7% of all under-five deaths in Kenya. Recent experiences in other countries show that the private health sector can be successfully harnessed to improve diarrhoea treatment coverage.

This study assesses the effect of prompting the supply of zinc and low-osmolarity oral rehydration salts (LO-ORS) co-packs in the private sector coupled with increasing the demand for co-packs among caregivers on: 1) the treatment of uncomplicated childhood diarrhoea, 2) care-seeking in the private sector, and 3) availability of co-packs in the private sector.

The target population will be children under five years of age and their caregivers in Vihiga County. The study will use a effectiveness-implementation hybrid design with two arms: 1) children and caregivers from areas that receive the current standard of care and will be exposed to standard BCC and 2) children and caregivers from areas where the private sector component will be implemented and that will be exposed to a modified BCC. Two of the five existing sub-counties in Vihiga will be selected by convenience to be assigned to one of the two study arms. The selection will take into account geographical distance between the two sub-counties (i.e. maximizing the distance between the two counties to minimize cross-pollination between the two study groups), rural vs urban population, and number of operational community units and CHV in each sub-county. All private sector retailers within each sub-county will be identified with assistance from wholesalers. Retailers will be invited to participate in the study via sensitization meetings.

Baseline and endline assessments will be conducted at the household level to collect information on care-seeking practices, availability of the co-pack in the household, treatment of diarrhoea, and whether caregivers received information from shopkeepers on using the co-pack. Monitoring of process indicators will be conducted throughout the intervention period. The monitoring process will also be used to evaluate the adoption and feasibility of the implementation model. In addition, the endline survey will be used to evaluate the acceptability, adoption, and coverage of the implementation model.

ELIGIBILITY:
Inclusion criteria:

* All children under 5 years of age who live in the selected areas to be included in the study are eligible to participate. All children in area selected for the intervention will be exposed to the private sector component and the modified BCC.
* In addition, all private sites (shops, kiosks, chemists) in the intervention area will be eligible to participate in the study.

Exclusion criteria:

- None

Ages: 2 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1245 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-04-02 (Actual); Study Completion 2022-04-02 (Actual)

PRIMARY OUTCOMES:
Treatment of uncomplicated diarrhea | 12 months
  change in % of caregivers who use zinc and LO-ORS co-pack to treat uncomplicated childhood diarrhea at 12 months
Care-seeking in the private sector | 12 months
  Change in % of caregivers seek care for uncomplicated childhood diarrhea in the private sector at 12 months
Availability of zinc and LO-ORS co-pack in the private sector | 12 months
  Change in % of private retailers who have stock of zinc and LO-ORS co-pack at time of visit at 12 months
Acceptability of private sector | 1 month
  % private retailers who express intention to stock co-packs after sensitization and training.
Acceptability of caregivers | 12 months
  % caregivers who indicate preferred treatment for uncomplicated childhood diarrhea is co-pack.at 12 months
Adoption by private sector at month 1 | 1 month
  % private retailers who stock co-pack after 1 month
Adoption by private sector at month 2 | 2 months
  % private retailers who stock co-pack after 2 months
Adoption by private sector at month 3 | 3 months
  % private retailers who stock co-pack after 3 months
Adoption by private sector at month 4 | 4 months
  % private retailers who stock co-pack after 4 months
Adoption by private sector at month 5 | 5 months
  % private retailers who stock co-pack after 5 months
Adoption by private sector at month 6 | 6 months
  % private retailers who stock co-pack after 6 months
Adoption by private sector at month 7 | 7 months
  % private retailers who stock co-pack after 7 months
Adoption by private sector at month 8 | 8 months
  % private retailers who stock co-pack after 8 months
Adoption by private sector at month 9 | 9 months
  % private retailers who stock co-pack after 9 months
Adoption by private sector at month 10 | 10 months
  % private retailers who stock co-pack after 10 months
Adoption by private sector at month 11 | 11 months
  % private retailers who stock co-pack after 11 months
Adoption by private sector at month 12 | 12 months
  % private retailers who stock co-pack after 12 months
Adoption by caregivers | 12 months
  % caregivers who indicate having co-pack in house
Feasibility of intervention at month 1 | 1 month
  % private retailers who indicate that they can purchase/procure co-packs with ease after 1 month
Feasibility of intervention at month 2 | 2 months
  % private retailers who indicate that they can purchase/procure co-packs with ease after 2 months
Feasibility of intervention at month 3 | 3 months
  % private retailers who indicate that they can purchase/procure co-packs with ease after 3 months
Feasibility of intervention at month 4 | 4 months
  % private retailers who indicate that they can purchase/procure co-packs with ease after 4 months
Feasibility of intervention at month 5 | 5 months
  % private retailers who indicate that they can purchase/procure co-packs with ease after 5 months
Feasibility of intervention at month 6 | 6 months
  % private retailers who indicate that they can purchase/procure co-packs with ease after 6 months
Feasibility of intervention at month 7 | 7 months
  % private retailers who indicate that they can purchase/procure co-packs with ease after 7 months
Feasibility of intervention at month 8 | 8 months
  % private retailers who indicate that they can purchase/procure co-packs with ease after 8 months
Feasibility of intervention at month 9 | 9 months
  % private retailers who indicate that they can purchase/procure co-packs with ease after 9 months
Feasibility of intervention at month 10 | 10 months
  % private retailers who indicate that they can purchase/procure co-packs with ease after 10 months
Feasibility of intervention at month 11 | 11 months
  % private retailers who indicate that they can purchase/procure co-packs with ease after 11 months
Feasibility of intervention at month 12 | 12 months
  % private retailers who indicate that they can purchase/procure co-packs with ease after 12 months

SECONDARY OUTCOMES:
Care-seeking to all sources | 12 months
  Change in % of caregivers who seek care for childhood diarrhea outside the home at month 12
Prompt treatment of uncomplicated childhood diarrhoea with zinc and LO-ORS co-pack | 12 months
  Change in % of caregivers who use zinc and LO-ORS co-pack to treat uncomplicated childhood diarrhea within 24-h of the onset of the episode of diarrhea at 12 months
Caregivers receive information from private retailers | 12 months
  Change in % caregivers who indicate received information from private retailers about zinc and LO-ORS to treat uncomplicated childhood diarrhea at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Elijah Mbiti, MSc, Principal Investigator — Nutrition International
Locations (1):
- Nutrition International - Kenya, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] United Nations Inter-agency Group for Child Mortality Estimation (UN IGME), 'Levels & Trends in Child Mortality: Report 2019, Estimates developed by the United Nations Inter-agency Group for Child Mortality Estimation', United Nations Children's Fund, New York, 2019
- [Background] GBD 2016 Diarrhoeal Disease Collaborators. Estimates of the global, regional, and national morbidity, mortality, and aetiologies of diarrhoea in 195 countries: a systematic analysis for the Global Burden of Disease Study 2016. Lancet Infect Dis. 2018 Nov;18(11):1211-1228. doi: 10.1016/S1473-3099(18)30362-1. Epub 2018 Sep 19. PMID 30243583
- [Background] UNICEF. Diarrhoeal disease - UNICEF DATA. 2018. Available from: https://data.unicef.org/topic/child-health/diarrhoeal-disease. (Accessed 24 Sept 2019)
- [Background] KDHS, Kenya Demographic and Health Survey. Kenya National Bureau of Statistics, the National AIDS Control Council (NACC), the National Council for Population and Development (NCPD), and the Kenya Medical Research Institute (KEMRI), ICF International. 2014.
- [Background] Walker CL, Black RE. Zinc for the treatment of diarrhoea: effect on diarrhoea morbidity, mortality and incidence of future episodes. Int J Epidemiol. 2010 Apr;39 Suppl 1(Suppl 1):i63-9. doi: 10.1093/ije/dyq023. PMID 20348128
- [Background] Munos MK, Walker CL, Black RE. The effect of oral rehydration solution and recommended home fluids on diarrhoea mortality. Int J Epidemiol. 2010 Apr;39 Suppl 1(Suppl 1):i75-87. doi: 10.1093/ije/dyq025. PMID 20348131
- [Background] International Vaccine Access Center (IVAC), Johns Hopkins Bloomberg School of Public Health. Pneumonia and Diarrhoea Progress Report 2015: Sustainable Progress in the Post-2015 Era. 2015.
- [Background] World Health Organization. Clinical Management of acute diarrhoea: WHO/UNICEF joint statement. 2004. Available: http://www.who.int/iris/handle/10665/68627. Accessed: 24 September 2019
- [Background] International Vaccine Access Center, Johns Hopkins Bloomberg School of Public Health. Pneumonia and Diarrhea Progress Report 2017: Pushing Progress through Investment & Action; 2017. Available from: https://www.jhsph.edu/research/centers-and-institutes/ivac/resources/IVAC-2017-Pneumonia-Diarrhea-Progress-Report.pdf. Accessed: 23 Sept 2019.
- [Background] Bradley, Sarah E. K., Lauren Rosapep, and Tess Shiras. 2018. Sources for Sick Child Care in Kenya. Brief. Rockville, MD: Sustaining Health Outcomes through the Private Sector Plus Project, Abt Associates
- [Background] ACTwatch Group. (2015). ACTwatch Outlet Surveys 2013-2014 - ORS and Zinc Availability Findings from 9 Countries. Washington DC: PSI.
- [Background] Kim Y, Hahn S, Garner P. Reduced osmolarity oral rehydration solution for treating dehydration caused by acute diarrhoea in children. Cochrane Database Syst Rev. 2001;2002(2):CD002847. doi: 10.1002/14651858.CD002847. PMID 11406049
- [Background] Lazzerini M, Wanzira H. Oral zinc for treating diarrhoea in children. Cochrane Database Syst Rev. 2016 Dec 20;12(12):CD005436. doi: 10.1002/14651858.CD005436.pub5. PMID 27996088
- [Background] Lamberti LM, Fischer Walker CL, Taneja S, Mazumder S, Black RE. The Association between Provider Practice and Knowledge of ORS and Zinc Supplementation for the Treatment of Childhood Diarrhea in Bihar, Gujarat and Uttar Pradesh, India: A Multi-Site Cross-Sectional Study. PLoS One. 2015 Jun 22;10(6):e0130845. doi: 10.1371/journal.pone.0130845. eCollection 2015. PMID 26098305
- [Background] Carter E, Bryce J, Perin J, Newby H. Harmful practices in the management of childhood diarrhea in low- and middle-income countries: a systematic review. BMC Public Health. 2015 Aug 18;15:788. doi: 10.1186/s12889-015-2127-1. PMID 26282400
- [Background] Goh N, Pollak K. Progress over a decade of zinc and ORS scale-up: Best practices and lessons learned. 2016. Available: https://www.defeatdd.org/reports/progress-over-decade-zinc-and-ors-scale. Accessed: 25 September 2019
- [Background] Data on policies, systems and financing. Countdown 2030 Master Databases (December 2017 Country Profiles). Countdown to 2030, Women's, Children's and Adolescents' Health. Available from: http://countdown2030.org/country-and-regional-networks/country-profiles/countdown-2030-master-databases-january-2018-country-profiles. Accessed: 23 September 2019
- [Background] Ministry of Public Health and Sanitation (2010). Policy Guidelines on control and Management of Diarrhoeal disease in Children below five years in Kenya. Nairobi.
- [Background] Ministry of Medical Services and Ministry of Public Health & Sanitation, (2010).Kenya Essential Medicines List 2010. Available at: http://apps.who.int/medicinedocs/documents/s18694en/s18694en.pdf. Accessed: 24 September 2019.
- [Background] Ministry of Health - Government of Kenya. (2016). Kenya Reproductive Maternal Newborn Child and Adolescent Health (RMNCHA) Investment Framework. Nairobi: Ministry of Health - Government of Kenya
- [Background] Ministry of Medical Services and Ministry of Public Health & Sanitation, (2016).Kenya Essential Medicines List 2016. Available at: http://apps.who.int/medicinedocs/documents/s23035en/s23035en.pdf. Accessed 24 Sept 2019.
- [Background] Every Women Every Child. 2012. UN Commission on life-savig commodities for women and children: commisioners' report. Available at: https://www.unicef.org/media/files/UN_Commission_Report_September_2012_Final.pdf. Accessed 24 Sept 2019
- [Background] Bedford KJ, Sharkey AB. Local barriers and solutions to improve care-seeking for childhood pneumonia, diarrhoea and malaria in Kenya, Nigeria and Niger: a qualitative study. PLoS One. 2014 Jun 27;9(6):e100038. doi: 10.1371/journal.pone.0100038. eCollection 2014. PMID 24971642
- [Background] Ahs J. Perceptions, Management and Barriers to Care-seeking for Childhood Diarrhea, Malaria, and Pneumonia: Uganda, Kenya, Nigeria, Ethiopia, Niger. 2012. North Carolina. USA
- [Background] ICF, 2012. The DHS Program STATcompiler. Funded by USAID. Available at: http://www.statcompiler.com. Accessed 24 Sept 2019.
- [Background] Kruger C, Heinzel-Gutenbrunner M, Ali M. Adherence to the integrated management of childhood illness guidelines in Namibia, Kenya, Tanzania and Uganda: evidence from the national service provision assessment surveys. BMC Health Serv Res. 2017 Dec 13;17(1):822. doi: 10.1186/s12913-017-2781-3. PMID 29237494
- [Background] Ross-Degnan D, Soumerai SB, Goel PK, Bates J, Makhulo J, Dondi N, Sutoto, Adi D, Ferraz-Tabor L, Hogan R. The impact of face-to-face educational outreach on diarrhoea treatment in pharmacies. Health Policy Plan. 1996 Sep;11(3):308-18. doi: 10.1093/heapol/11.3.308. PMID 10160376
- [Background] NCAPD, MOMS, MOPHS, KNBS, ICF Macro. (2011). Kenya Service Provision Assessment Survey 2010. Nairobi, Kenya: National Coordinating Agency for Population and Development, Ministry of Medical Services, Ministry of Public Health and Sanitation, Kenya National Bureau of Statistics, and ICF Macro.
- [Background] UNICEF Supply Division. Oral Rehydration Salts and Zinc: UNICEF Suppliers and Product Range. February 2016. Availabel at: https://www.unicef.org/supply/files/ORS_and_Zinc_Supply_Update_1_-_with_warning_banner.pdf. Accessed: 24 Sept 2019.
- [Background] Larson CP, Saha UR, Nazrul H. Impact monitoring of the national scale up of zinc treatment for childhood diarrhea in Bangladesh: repeat ecologic surveys. PLoS Med. 2009 Nov;6(11):e1000175. doi: 10.1371/journal.pmed.1000175. Epub 2009 Nov 3. PMID 19888335
- [Background] Larson CP, Koehlmoos TP, Sack DA; Scaling Up of Zinc for Young Children (SUZY) Project Team. Scaling up zinc treatment of childhood diarrhoea in Bangladesh: theoretical and practical considerations guiding the SUZY Project. Health Policy Plan. 2012 Mar;27(2):102-14. doi: 10.1093/heapol/czr015. Epub 2011 Feb 22. PMID 21343236
- [Background] SHOPS. Increasing the Use of ORS and Zinc through the Private Sector. 2018. Available at: https://www.shopsplusproject.org/sites/default/files/resources/Zinc_Final_.pdf. Accessed 24 Sept 2019.